CLINICAL TRIAL: NCT00957489
Title: A Prospective Randomized Controlled Trial to Evaluate the Effectiveness of the Two Different Appliances in the Treatment of Class II Division 1 Malocclusion
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study stopped due to increased harm and slow progress in the intervention group.
Sponsor: University of Manchester (Other)
Collaborators: National Health Service, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Badri Thiruvenkatachari, Dr, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DTT project
Record Dates: First submitted 2009-08-11; First posted 2009-08-12 (Estimated); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Class II Division 1 Malocclusion
Keywords: Orthodontic treatment of Class II division 1 malocclusion
MeSH Terms: conditions — Malocclusion, Angle Class II

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Functional appliance-Dynamax (Experimental)
  Interventions: Other: Dynamax appliance
- Functional appliance- twin block (Other): Conventional treatment
  Interventions: Other: Twin-block appliance

INTERVENTIONS:
Other: Dynamax appliance
  Arms: Functional appliance-Dynamax
Other: Twin-block appliance
  Arms: Functional appliance- twin block

SUMMARY:
Twin-Block treatment and Dynamax treatment for Class II division 1 malocclusion do not have different effects with regards to treatment duration, the quality of dento-occlusal outcome, skeletal and soft tissue profile, patient discomfort and gingival health.

DETAILED DESCRIPTION:
The Dynamax appliance is a relatively new appliance for the treatment of Class II malocclusion and was introduced in 2003. The appliance has the theoretical advantages of incremental mandibular advancement without the need for bite registration, and the ability for the operator to simultaneously provide the functional and fixed appliance phases of treatment. Furthermore, the Dynamax appliance is designed to limit lower both lower incisor proclination and upper incisor retroclination without an increase in lower facial height. There has been limited research into this appliance and only one trial has been carried out. In this study the effects of the Dynamax were compared with the Twin-block, unfortunately, the trial was not carried out to contemporary standards and suffered from severe shortcomings. For example, the non compliance rate was not accounted for in the sample size calculation, the randomisation sequence was not clear, the investigators did not carry out an intention-to-treat analysis, the statistical analysis was simplistic and the study was carried out in a single dental school setting. This raises the question about the efficiency of the Dynamax appliance and whether or not they are effective in a 'real' world setting.

The aim of this study is to compare the effectiveness of the Dynamax appliance and the Twin-block appliance for the treatment of Class II Division 1 malocclusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a Class II malocclusion as defined by British Standards Institute classification.
* Overjet greater than 6mm
* Aged 10-14 years
* Clinical examination indicates a functional appliance is not contraindicated

Exclusion Criteria:

* Orthognathic treatment is required or there is a strong indication it will be required in the future
* Possession of a craniofacial anomaly
* Previous orthodontic treatment and/or premolar extraction
* Hypodontia of more than one teeth in any quadrant excluding third molars
* Inadequate oral hygiene

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2007-01; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Duration of treatment with functional appliance | 9 months
Overjet measurement | 9 months

SECONDARY OUTCOMES:
Harms Breakages Number of treatment visits Total treatment time Quality of occlusal result (PAR Index) Restricted cephalometric (radiograph) analysis Patient perception questionnaire at six months into treatment | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Kevin O'Brien, BDS, MSc, FDSRCS, DORth, PhD, Principal Investigator — Prof of Orthodontics/ Associate Dean Teaching and Learning, University of Manchester; Jonathan Sandler, BDS, MSc, FDSRCS, MOrth RCS, Principal Investigator — Consultant Orthodontist, Chesterfield NHS Trust; Alison Murray, BDS, MSc, FDSRCS, MORth RCS, Principal Investigator — Consultant Orthodontist, Derby NHS Trust; Badri ' Thiruvenkatachari, BDS, MDS, MOrth RCS, PhD, Study Director — Clinical Teaching Fellow in Orthodontics, University of Manchester
Locations (2):
- United Kingdom (2):
  - Chesterfield Royal Hospital, Chesterfield
  - Derby Royak Hospital NHS Trust, Derby